CLINICAL TRIAL: NCT02721251
Title: Influence of Exercise, Weight Loss, and Exercise Plus Weight Loss on Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Behind enrollment targets
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNB-012-14S
Record Dates: First submitted 2016-02-17; First posted 2016-03-29 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Sleep Apnea; Overweight
Keywords: exercise; weight loss; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Overweight; Motor Activity; Weight Loss; Sleep Apnea Syndromes | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise (Experimental): 16 week intervention, building up to 30-45 minutes of aerobic exercise 4 days per week, and 15 min of resistance exercise 2 days per week
  Interventions: Behavioral: Exercise
- Weight Loss (Experimental): 16 week intervention with a goal weight loss of 10%, accomplished with caloric and fat restriction, weekly sessions with a nutritionist, and some meal replacement
  Interventions: Behavioral: Weight Loss
- Exercise + Weight Loss (Experimental): Combined components of the exercise and weight loss treatments
  Interventions: Behavioral: Exercise + Weight Loss

INTERVENTIONS:
Behavioral: Exercise — 16 weeks. 4 days per week of aerobic exercise; 45 min for 2 days and for 30 min for two days. 2 days per week of resistance exercise for 15 min (coinciding with the days involving 30 min of aerobic exercise)
  Arms: Exercise
Behavioral: Weight Loss — 16 week. the goal is 10% weight loss.
  Arms: Weight Loss
Behavioral: Exercise + Weight Loss — Combined exercise and weight loss components of the other arms
  Arms: Exercise + Weight Loss

SUMMARY:
Obstructive sleep apnea (OSA) is highly prevalent among Veterans, and is associated with significant mortality and multiple morbidities. Available treatments have had limited effectiveness in treating OSA and alleviating associated morbidity. The investigators' previous research found a reduction in OSA severity of approximately 25% following modest exercise training. That this effect occurred independent of weight loss raises the exciting possibility that exercise combined with weight loss could reduce OSA by at least 50% and have unique health benefits for OSA patients. Following screening and baseline assessments, 90 overweight Veterans ages 18-60 years with OSA will be randomized to one of three 16-week treatments: (1) exercise training; (2) 10 % weight loss; and 3) exercise + weight loss. Changes in OSA and related morbidity will be compared between treatments.

DETAILED DESCRIPTION:
Rationale: Approximately 15-20% of adults have obstructive sleep apnea (OSA), and evidence indicates that the prevalence of OSA is perhaps twice as high among Veterans. OSA has been clearly linked to increased mortality and multiple morbidities, and undoubtedly contributes to the high prevalence of health problems among Veterans. Current treatments for OSA are not well tolerated, often have limited efficacy, and often do not result in improvements in health. The investigators' recent research demonstrated that 12 weeks of moderate exercise training elicited a reduction of OSA of ~25%, as well as significant improvement in mood, fatigue, quality of life, and cardiovascular health. Interestingly, as with other health benefits of exercise, the investigators' research is consistent with other research showing that exercise can reduce OSA independent of changes in body weight. These studies raise the exciting possibility that exercise training combined with modest weight loss could elicit a chronic reduction in OSA of 50% or more.

Objectives: The investigators' Objective is to compare the effects of 16 weeks of exercise training alone, weight loss alone, and exercise + weight loss on OSA severity and associated morbidity.

Methods: Following extensive screening and baseline assessment, N=90 overweight/obese Veterans (ages 18-60 years) with mild to severe OSA will be randomized to one of three 16-week treatments. (1) Exercise Alone (n=30) will involve training 4 days per week under supervision of a clinical exercise physiologist. It will include aerobic exercise (treadmill, cycling, elliptical) that will gradually increase to 30-45 min on 4 days/wk, as well as resistance exercise (15 min) on 2 days/week. (2) Weight Loss Alone (n=30) will involve a structured meal plan (including some meal replacement with shakes or bars), and weekly counseling designed to elicit a reduction in body weight of 10%. (3) Exercise + Weight Loss (n=30) will involve the same exercise and weight loss interventions as in the other treatments. Outside of the interventions, participants will be asked to maintain their usual exercise and diet habits, as verified, respectively, with actigraphic recording and a 24-hr food recall. Before and after the treatments, participants will undergo 5 days/nights of home-based actigraphic and diary-assessed sleep, and one night of laboratory polysomnographic recording of sleep, including OSA severity. Comorbidity measures will include pre- to post-treatment changes in blood pressure, glucose, insulin, lipids, hemoglobin a1c, body weight/composition, and inflammation (e.g., CRP, IL-6). Also measured will be monthly changes in self-reports of sleep quality, functional outcomes of sleepiness (FOSQ), and snoring symptoms. A 3-month follow-up will include home assessment of OSA, as well as sleep quality, FOSQ, and snoring. Mediation analysis will explore whether improvements in OSA are mediated by changes in percent of deep sleep, body weight, trunk body fat percent, trunk total mass, respiratory muscle strength, and upper airway obstruction assessed in the laboratory.

Implications for Future Research. Demonstration of a reduction of OSA by 50% would result in extensive subsequent studies. These would likely include studies of dose-response effects; comparisons of different modes of exercise; studies of the feasibility of telemedicine approaches to the interventions; comparative efficacy studies vs. PAP; further mechanistic studies, for example, of upper airway collapsibility and composition (e.g, via MRI); and studies of other positive health outcomes, such as extensive heart imaging.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* 18-65 years of age
* Moderate-severity OSA [[Apnea-hypopnea index (AHI) 15 at screening]
* Overweight/obese
* Physically inactive
* BMI 28
* Sedentary lifestyle (planned activity for purpose of health < 2 days/week)
* Stable weight Not engaged in weight loss study or program
* Stable medications Medications for thyroid, cholesterol, blood pressure, and other conditions at same dose for 2 months
* Capable of signing consent and willing to provide informed consent and accept randomization assignment

Exclusion Criteria:

* Current OSA treatment Current use of continuous positive airway pressure (PAP), dental devices, etc. for OSA treatment. Past PAP or oral appliances are not exclusions if discontinued 2 months before study
* Significant disease: known or signs/symptoms of cardiovascular, metabolic, or pulmonary disease
* Uncontrolled hypertension: Blood pressure > 159/99 mmHg
* Unable to exercise: musculoskeletal, orthopedic, neuromuscular, or other conditions that do not allow exercise or where exercise is contraindicated
* Any accident attributable to sleepiness in previous 3 years
* Current pregnancy/planning to become pregnant
* Clinically judged unsuitable as evaluated by supervising medical physician

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D. Youngstedt, PhD, Principal Investigator — Phoenix VA Health Care System, Phoenix, AZ
Locations (1):
- Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 signed consent. Of these, 31 did not pass screening for various reasons, and 5 participants were not able to complete screening procedures after the study was stopped. Thus, 47 participants were randomized to one of the three treatments
Pre-assignment Details: Reasons for not passing screening procedures for various reasons, including insufficiently severe sleep apnea. Of the 47 participants who started one of the treatments, 24 dropped out during the study, for various reasons, including burden of the intervention, transportation difficulties, going to jail. Six other participants were excluded for non-adherence. Thus, 17 participants completed the study.
Period: Overall Study
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Started | 14 | 16 | 17
Completed | 4 | 7 | 6
Not Completed | 10 | 9 | 11
Not completed — Withdrawal by Subject | 8 | 7 | 9
Not completed — poor adherence | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Information on those who started the intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss | Total
Number analyzed (Participants) | 14 | 16 | 17 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 17 | 47
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (10.3) | 49.1 (9.7) | 48.2 (8.5) | 49.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 13 | 15 | 15 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 6
  Not Hispanic or Latino | 13 | 13 | 15 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 8
  White | 9 | 10 | 13 | 32
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI)
Description: Common criterion for obstructive sleep apnea: number of apnea and hypopnea episodes per hour of sleep. Baseline-end - positive value indicates a reduction.
Time Frame: Change from baseline to the end of the study (16-week intervention)
Population: Data on the final AHI are missing for one participants in the exercise + weight loss treatment.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Weight Loss: 16 week intervention with a goal weight loss of 10%, accomplished with caloric and fat restriction, weekly sessions with a nutritionist, and some meal replacement Weight Loss: 16 week. the goal is 10% weight loss.
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 4 | 7 | 5
events per hour | 17.8 (26.9) | -4.3 (8.7) | -10.7 (7.0)

2. Secondary Outcome: Functional Outcomes of Sleepiness Questionnaire (FOSQ)
Description: Measures impairments in functioning associated with sleepiness. Baseline minus end of study value. Positive value indicates improvement; negative value indicates worsening.
  Minimum score on scale: 0 Maximum score: 120
Time Frame: Change from baseline to the end of the study (16-week intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 4 | 7 | 6
units on a scale | -22.7 (14.1) | -13.6 (19.1) | -0.33 (41.0)

3. Secondary Outcome: Snoring Severity Scale
Description: Questionnaire that measures severity of snoring with a questionnaire. A positive value indicates improvement; a negative value indicates worsening.
  Minimum score: 0 Maximum score: 9
Time Frame: Change from baseline to the end of the study (16-week intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 4 | 7 | 6
units on a scale | 2.3 (3.9) | 1.0 (2.2) | 0.3 (2.9)

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Commonly used metric of sleep quality. Baseline minus end of study. Positive value indicates improvement.
  Minimum score: 0 Maximum score: 21
Time Frame: Change from baseline to the end of the study (16-week intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 4 | 7 | 6
units on a scale | 0.9 (0.6) | -0.7 (0.6) | 1.0 (2.6)

5. Secondary Outcome: Blood Pressure
Description: Blood pressure
Time Frame: Change from baseline to the end of the study (16-week intervention)
Population: Data missing
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Body Weight
Description: Fasting body weight. Weight change (kg) beginning to end of study (positive valuate = decrease)
Time Frame: Change from baseline to the end of the study (16-week intervention)
Population: Final body weight data are missing on n=1, 3, and 2 participants in the weight loss, exercise, and exercise + weight loss treatment, respectively.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 3 | 4 | 4
kg | 5.0 (6.9) | 0.2 (4.7) | 8.0 (10.3)

7. Secondary Outcome: Percent Body Fat Assessed With Dual-energy X-reay Absorptiometry (DEXA)
Description: Percent body fat assessed with DEXA. Change in percent body fat - positive value represents a decrease.
Time Frame: Change from baseline to the end of the study (16-week intervention)
Population: Data are missing for n=2, 3, and 2 participants in the weight loss, exercise, and exercise + weight loss treatments, respectively.
Measure: Mean (Standard Deviation); unit: change in % body fat
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 2 | 4 | 4
change in % body fat | 0.6 (0.4) | 0.8 (0.9) | 1.6 (0.3)

8. Secondary Outcome: C-reactive Protein (CRP)
Description: Measure of inflammation
Time Frame: Change from baseline to the end of the study (16-week intervention)
Population: Unable to locate data
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: VA procedures
Arm/Group | Weight Loss | Exercise | Exercise + Weight Loss
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02721251/Prot_SAP_000.pdf